CLINICAL TRIAL: NCT03135041
Title: Effects of a Combination of Prebiotic Fibres on Weight Loss During an Energy Restricted Diet in an Overweight/Obese Population
Brief Title: The Effect of Prebiotic Fibres on Weight Loss in an Overweight and Obese Population
Acronym: MNGII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Reading (Other); TNO (Other); National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Thomas Meinert Larsen, Associate Professor, PhD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B328
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Prebiotics; Microbiome; Glucose metabolism
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber-containing dietary supplement (Experimental): 2 x 200 ml of fiber-enriched UHT milk during 12 weeks of energy restriction
  Interventions: Dietary Supplement: Fiber-containing dietary supplement
- Placebo (Placebo Comparator): 2 x 200 ml of UHT milk with maltodextrin during 12 weeks of energy restriction
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fiber-containing dietary supplement — Effects of fiber-containing dietary supplement on weight loss during energy restriction
  Arms: Fiber-containing dietary supplement
Dietary Supplement: Placebo — Effects of placebo supplement on weight loss during energy restriction
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether a diet supplemented with two prebiotic fibres induces greater changes in body weight compared to placebo during 12 weeks of energy restriction in an obese/overweight population.

The hypothesis is that the fiber-containing dietary supplement will:

1) Induce greater changes in body weight compared to the placebo group 2) change the gut microbiota composition 3) improve glucose homeostasis 4) decrease serum concentration of triglycerides, total and LDL cholesterol

The hypothesis is that the effect of the intervention on weight loss will be partly mediated by the diet-induced changes in the gut microbiota composition.

DETAILED DESCRIPTION:
Prebiotics are nutrients that specifically utilized by the gut microbiota. Beneficial health effects of prebiotics are generally attributed to 1) stimulation of beneficial bacteria and SCFA production, and consequently; improved barrier function, regulation of enteroendocrine peptide secretion and resistance to inflammatory stimuli; 2) modulation of lipid metabolism, possibly by suppression of lipogenic enzymes and thus decreased synthesis of lipoproteins and triglycerides; and 3) increased mineral absorption.

Inulin is recognized as a common prebiotic. Fibersol-2 is a resistant starch that has been suggested to induce satiety, when given in a dose of 10 g. Intake of inulin has been shown to induce changes in the microbial abundance and increase production of SCFA19; whereas resistant starch has been shown to improve insulin sensitivity and postprandial glucose AUC20. However, the effects of an intervention with a combination of these two fibers on obesity and body composition during an energy restricted diet have not been addressed. Supplements with other types of fibres in addition to energy restriction have shown additional effects in weight reduction.

In this study, the effects of a combination product of two prebiotic fibres on additional weight loss during energy restriction in a placebo-controlled, randomized parallel study with a duration of 12 weeks will be tested. Furthermore, the effects of the fibres on the gut microbial composition, markers of metabolic syndrome (MetS) and glucose metabolism will be tested. The active diet will contain intervention products high in dietary fibre and the placebo diet will contain maltodextrin. The fiber-containing dietary supplements will add approximately 20 g of prebiotic fibres per day, where approximately 10 g will be inulin and approximately 10 g will be resistant maltodextrin. The intervention products and placebo will be consumed as milk. The fiber-containing dietary supplement is expected to induce additional weight loss, compared to placebo and to affect the gut microbiome and markers of metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 28-45 kg/m2
* Non-smoking
* Haemoglobin level ≥7 mmol/L

Exclusion Criteria:

* Use of antibiotics three months prior to study and during the study. If a participant uses antibiotics prior to randomization, the participant will be invited to be re-screened 3 months after the last use of antibiotics, provided that it is realistic to complete the study no later than the scheduled LPLV
* Weight change >3 kg two months prior to study
* Blood donation other than for this study <1 month prior to study and during study.
* Participation in clinical trials other than for this <1 month prior to study and during study
* Intensive physical training/ elite athlete (>10 hours of strenuous physical activity per week)
* Unstable medication for dyslipidaemia and elevated blood pressure (the participant must have had a stable dose in the three months prior to study start), and use of systemic glucocorticoids
* Medication for T2D
* Treatment with metformin
* Dietary supplements with pro- and/or prebiotics and/or fibre 6 weeks prior to study
* Special dietary regimen (vegetarians, vegans etc.), as evaluated by study staff
* Lactose intolerance or allergy to components in the intervention products
* Gluten intolerance
* Maltodextrin intolerance
* Lactation, pregnancy or planning of pregnancy during the study
* Gastro intestinal and liver disorders
* Chronic inflammation disorders (excluding obesity)
* Diagnosed psychiatric disorder including depression requiring treatment
* Surgical treatment of obesity and abdominal surgery
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the study staff

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Weight loss | Measurements will be performed at baseline and after 12 weeks of intervention
  Differences in changes in body weight between the group that receives fiber-containing dietary supplement and placebo group

SECONDARY OUTCOMES:
Body composition | Measurements will be performed at baseline and after 12 weeks of intervention
  Changes in body composition
Gut microbiota composition and function | Measurements will be performed at baseline and after 12 weeks of intervention
  Changes in gut microbiota composition and function (faecal samples) assesed by metagenomics
Glucose metabolism | Measurements will be performed at baseline and after 12 weeks of intervention
  Glucose and insulin homeostasis
Lipid metabolism | Measurements will be performed at baseline and after 12 weeks of intervention
  Analyses of lipids in blood samples
Inflammatory markers | Measurements will be performed at baseline and after 12 weeks of intervention
  Changes in concentration of inflammatory markers
SCFA concentration | Measurements will be performed at baseline and after 12 weeks of intervention
  Changes in faecal concentration of short chain fatty acids
Lipidomics and bile acids | Measurements will be performed at baseline and after 12 weeks of intervention
  Changes in concentration of lipids and bile acids in blood and faecal samples
Metabolomics | Measurements will be performed at baseline and after 12 weeks of intervention
  Analyses of metabolites in blood, urine and fecal samples
Weight loss | Measurements will be performed at baseline and after 12 weeks of intervention
  Interaction between differences in changes in body weight between the group that receives fiber-containing dietary supplement and placebo group and each of baseline fasting glucose, baseline fasting insulin and baseline microbiome composition (e.g. enterotype).

OTHER OUTCOMES:
Physical activity | Measurements will be performed at baseline and after 12 weeks of intervention
  Measurement of physical activity, as assessed by Actigraph monitors
Appetite regulation | Measurements will be performed at baseline and after 12 weeks of intervention
  Markers of appetite regulation
Gene expression | Measurements will be performed at baseline and after 12 weeks of intervention
  Measurements of gene expression in of selected genes
Epigenetics | Measurements will be performed at baseline and after 12 weeks of intervention
  Measurements of epigenetic markers in biological samples
Blood pressure | Measurements will be performed at baseline and after 12 weeks of intervention
  Blood pressure measured by an automated blood pressure monitor
Liver markers | Measurements will be performed at baseline and after 12 weeks of intervention
  Measurement of markers of liver health

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Larsen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Shared personal data collected includes basic data and demographics as well as health related data (weight, blood pressure, medical history etc.) and biological samples including maximum 50 mL blood, faecal samples and spot urine collected at baseline and during the study. The blood samples collected will be used for the analyses of markers of glucose metabolism, lipid metabo-lism and inflammation. Urine collection will be used for metabolomics analyses. Faecal samples will be used for metagenomics analyses and analysis of bile acids. Biological samples will be stored in the research biobank for 5 years and destroyed afterwards.
  Link between participant number and personal identification will be separated and stored in one protected participant number log.
  Personal data will be stored for 5 years, where data will be anonymized by destroying basic data sheet and participant number log.

REFERENCES:
- [Derived] Hess AL, Benitez-Paez A, Blaedel T, Larsen LH, Iglesias JR, Madera C, Sanz Y, Larsen TM; MyNewGut Consortium. The effect of inulin and resistant maltodextrin on weight loss during energy restriction: a randomised, placebo-controlled, double-blinded intervention. Eur J Nutr. 2020 Sep;59(6):2507-2524. doi: 10.1007/s00394-019-02099-x. Epub 2019 Oct 11. PMID 31605197